CLINICAL TRIAL: NCT01697111
Title: A Multi-center, Randomized, Double-blinded, Placebo-controlled, and Open-label, Active-controlled, Parallel-group Comparative Study to Assess Efficacy and Safety of an Extended Flexible Regimen of BAY 86-5300 [0.02 mg Ethinylestradiol (β-CDC) and 3 mg Drospirenone] in the Patients With Endometriosis
Brief Title: Comparative Study of BAY86-5300 With an Extended Flexible Regimen for Endometriosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15457
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-01

CONDITIONS: Endometriosis
Keywords: YAZ; Flexible regimen; Drospirenone; Ethinylestradiol Betadex; Endometriosis; Dienogest; Japanese Patients
MeSH Terms: conditions — Endometriosis | interventions — dienogest

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: EE20/DRSP(BAY86-5300)
- Arm 2 (Experimental)
  Interventions: Drug: Placebo
- Arm 3 (Active Comparator)
  Interventions: Drug: Dienogest

INTERVENTIONS:
Drug: EE20/DRSP(BAY86-5300) — One tablet [0.02 mg of ethinylestradiol (β-CDC) and 3 mg of drospirenone] / day
  Arms: Arm 1
Drug: Placebo — One tablet (no active ingredient) / day and one tablet [0.02 mg of ethinylestradiol (β-CDC) and 3 mg of drospirenone] / day, for the first 24 weeks and the later 28 weeks, respectively
  Arms: Arm 2
Drug: Dienogest — Dienogest 1mg twice a day (bid)
  Arms: Arm 3

SUMMARY:
This is a multi-center, randomized, double-blinded, placebo-controlled, parallel-group study (24-week treatment-comparison phase) with an open-label reference arm of active comparator (dienogest) followed by 28-week long-term treatment phase.

The primary objective of this study is to confirm the superiority of BAY86-5300 when administered with an extended flexible regimen for the treatment of endometriosis-associated pelvic pain in comparison to placebo in Japanese endometriosis patients within 24 weeks.

The secondary objective is to investigate the long-term safety of BAY86-5300 in patients treated with an extended flexible regimen for one year, and the bleeding pattern of BAY86-5300 when administered with an extended flexible regimen compared to dienogest.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as having endometriosis by laparotomy or laparoscopy, or by identification of chocolate cyst of endometriosis, or patients with the clinical diagnosis of endometriosis, who fulfill the condition of pelvic tenderness or induration of Cul-de-sac or uterine immobility
* Patient with pelvic pain judged by the highest Visual Analogue Scale (VAS) value of 40 mm or higher which is determined during 2 menstrual cycles before randomization (baseline observation phase)
* Patients having the normal menstrual cycle (25 to 38 days) in the latest two menses before randomization (baseline observation phase)
* Patients who do not wish to become pregnant during the course of the study

Exclusion Criteria:

* Patients who have organic diseases of which surgical treatment is prioritized by investigator
* Patients in whom any hormonal therapies, including combined oral contraceptives (COCs) and progestins, have failed for treatment of symptomatic endometriosis (moderate, severe pain)
* Patients for whom YAZ Combination Tablet is contraindicated (according to Japanese Labeling)
* Patients for whom dienogest is contraindicated (according to Japanese labeling of Dinagest Tab 1mg)

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2012-10; Primary Completion 2014-03 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change of pelvic pain from baseline period (8 weeks before start of treatment) to period of treatment (weeks 17-24) | Baseline period (8 weeks before start of treatment) and period of treatment (weeks 17-24)
  The pelvic pain is measured as the severest pain marked by the participant on a Visual Analogue Scale (VAS)

SECONDARY OUTCOMES:
Pelvic pain during menstrual or withdrawal bleeding period (except for dyspareunia and defecation pain) | Weeks 17-24 of treatment period
  Pelvic pain is the worst pain on a 0-10 scale rated by the participant.
Pelvic pain during non-menstrual period and non-withdrawal bleeding period (except for dyspareunia and defecation pain) | Weeks 17-24 of treatment period
  Pelvic pain is the worst pain on a 0-10 scale rated by the participant.
Dyspareunia | Weeks 17-24 of treatment period
  In case having sexual intercourse, dyspareunia pain is the worst pain on a 0-10 scale rated by the participant in the last 24 hours.
Average of pain | Weeks 17-24 of treatment period
  The average of pain is the mean value of the Visual Analogue Scale (VAS) value during the time frame calculated for each patient based on daily record of Patient Diary.
Size of chocolate cyst | 24 weeks after taking the initial study medication
  In case chocolate cyst is detected, size of chocolate cyst is a mean length (mm) of the longest axis and the short axis (crossing) of the largest chocolate cyst determined by transvaginal ultrasonography.
Endometrial thickness | 24 weeks after taking the initial study medication
  Endometrial thickness is the thickest value (mm) of endometrium determined by transvaginal ultrasonography.
Number of days with spotting/bleeding | Up to 52 weeks
  Number of days with spotting/bleeding is determined based on daily record of Patient Diary.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (25):
- Japan (25):
  - Anjo, Aichi-ken
  - Ichinomiya, Aichi-ken
  - Nagoya, Aichi-ken
  - Matsudo, Chiba
  - Fukui-shi, Fukui
  - Gifu, Gifu
  - Takasaki, Gunma
  - Itami, Hyōgo
  - Kawanishi, Hyōgo
  - Kobe, Hyōgo
  - Kanazawa, Ishikawa-ken
  - Kamakura, Kanagawa
  - Kawasaki, Kanagawa
  - Yokohama, Kanagawa
  - Osaka, Osaka
  - Toyonaka, Osaka
  - Kitamoto, Saitama
  - Bunkyo, Tokyo
  - Chuo-ku, Tokyo
  - Fuchū, Tokyo
  - Hachiōji, Tokyo
  - Machida, Tokyo
  - Minato, Tokyo
  - Nishitōkyō, Tokyo
  - tabashi City, Tokyo

REFERENCES:
- [Derived] Harada T, Kosaka S, Elliesen J, Yasuda M, Ito M, Momoeda M. Ethinylestradiol 20 mug/drospirenone 3 mg in a flexible extended regimen for the management of endometriosis-associated pelvic pain: a randomized controlled trial. Fertil Steril. 2017 Nov;108(5):798-805. doi: 10.1016/j.fertnstert.2017.07.1165. Epub 2017 Sep 11. PMID 28911925